CLINICAL TRIAL: NCT01230541
Title: Effect of Udenafil on Spermatogenesis: A Double-blind, Randomized, Placebo-controlled, Parallel-group Study
Brief Title: Effect of Udenafil on Spermatogenesis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: PR-00110
Record Dates: First submitted 2010-10-27; First posted 2010-10-29 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Spermatogenesis; Erectile Dysfunction
Keywords: Semen characteristics; Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — udenafil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Udenafil (Active Comparator): Udenafil daily tablet
  Interventions: Drug: Udenafil

INTERVENTIONS:
Drug: Placebo — Daily, oral tablet
  Arms: Placebo
Drug: Udenafil — Daily tablet
  Arms: Udenafil

SUMMARY:
Study of udenafil daily in subjects with mild or no erectile dysfunction to evaluate effects on semen characteristics.

DETAILED DESCRIPTION:
Safety Study in male subjects with no or mild ED (erectile dysfunction)

ELIGIBILITY:
Inclusion Criteria:

* No or mild ED (erectile dysfunction) willing & able to provide 2 semen samples without the use of PDE-5 inhibitor or other excluded medication or devices on 2 separate days during screening and at Weeks 12 & 26
* BMI (body mass index) between 19 and 31 kilogram/meter squared

Exclusion Criteria:

* New onset coronary artery disease within last 3 months, history of myocardial infarction or cardiac surgical procedure within last 6 months or sudden cardiac arrest
* Nitrate medications for angina pectoris
* Used of anti-arrhythmic drug treatment or device
* Congestive heart failure
* Uncontrolled diabetes
* Stroke or transient ischemic attack (TIA) within last 6 months
* Bleeding disorder or history of GI bleeding within last 12 months
* Cancer chemotherapy
* History of alcohol or drug abuse

Ages: 25 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 239 (Actual)
Dates: Start 2010-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Sperm Concentration Reduction greater than or equal to 50% at Week 26 | 26 weeks
  Percentage of Subjects with greater than or equal to 50% decrease from baseline in sperm concentration at 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Herman Ellman, MD, Study Director — Warner Chilcott
Locations (22):
- United States (22):
  - Warner Chilcott Investigational Site, Huntsville, Alabama
  - Warner Chilcott Investigational Site, Anaheim, California
  - Warner Chilcott Investigational Site, San Diego, California
  - Warner Chilcott Investigational Site, Tarzana, California
  - Warner Chilcott Investigational Site, Middlebury, Connecticut
  - Warner Chilcott Investigational Site, Aventura, Florida
  - Warner Chilcott Investigational Site, Clearwater, Florida
  - Warner Chilcott Investigational Site, Doral, Florida
  - Warner Chilcott Investigational Site, Ocala, Florida
  - Warner Chilcott Investigational Site, Pinellas Park, Florida
  - Warner Chilcott Investigational Site, Atlanta, Georgia
  - Warner Chilcott Investigational Site, Shreveport, Louisiana
  - Warner Chilcott Investigational Site, Plainsboro, New Jersey
  - Warner Chilcott Investigational Site, Garden City, New York
  - Warner Chilcott Investigational Site, Great Neck, New York
  - Warner Chilcott Investigational Site, Purchase, New York
  - Warner Chilcott Investigational Site, Williamsville, New York
  - Warner Chilcott Investigational Site, Cincinnati, Ohio
  - Warner Chilcott Investigational Site, San Antonio, Texas
  - Warner Chilcott Investigational Site, Webster, Texas
  - Warner Chilcott Investigational Site, Norfolk, Virginia
  - Warner Chilcott Investigational Site, Spokane, Washington